CLINICAL TRIAL: NCT02624401
Title: The Neural Mechanisms of Anesthesia and Human Consciousness (Part 6)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: University of California, Irvine (Other); University of Michigan (Other); Yale University (Other); University of Helsinki (Other)
Responsible Party: Principal Investigator, Harry Scheinin, Adjunct Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOC-2016
Record Dates: First submitted 2015-11-25; First posted 2015-12-08 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Anesthesia; Unconsciousness
MeSH Terms: conditions — Unconsciousness | interventions — Dexmedetomidine; Propofol; Esketamine; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dexmedetomidine (Experimental): Intravenous dexmedetomidine using target controlled infusion.
  Interventions: Drug: Dexmedetomidine
- Propofol (Experimental): Intravenous propofol using target controlled infusion.
  Interventions: Drug: Propofol
- S-ketamine (Experimental): Intravenous S-ketamine using target controlled infusion.
  Interventions: Drug: S-ketamine
- Sevoflurane (Experimental): Inhalational sevoflurane using target controlled inhalation.
  Interventions: Drug: Sevoflurane
- Placebo (Placebo Comparator): Intravenous saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous infusion
  Other Names: Dexdor
  Arms: Dexmedetomidine
Drug: Propofol — Intravenous infusion
  Other Names: Propofol-Lipuro
  Arms: Propofol
Drug: S-ketamine — Intravenous infusion
  Other Names: Ketanest-S
  Arms: S-ketamine
Drug: Sevoflurane — Inhalation
  Other Names: Sevorane
  Arms: Sevoflurane
Drug: Placebo — Intravenous infusion of saline (Ringer's Acetate)
  Arms: Placebo

SUMMARY:
Positron Emission Tomography (PET), Magnetic Resonance Imaging (MRI) and electroencephalography (EEG) studies will be carried out to reveal the neural correlates of consciousness. Consciousness of the subjects will be manipulated with anesthetic agents dexmedetomidine, propofol, S-ketamine and sevoflurane. One-hundred-and-sixty (160) healthy male subjects will be recruited to receive EC50 concentration of the anesthetic (40 dexmedetomidine, 40 propofol, 20 S-ketamine, 40 sevoflurane) or placebo (20) while being imaged for cerebral metabolic rate of glucose (CMRglu). Also genetic, immunological and metabolomics samples will be taken and analysed to find possible genetic factors explaining the variability in drug response and to find chemical fingerprints of acute drug effect.

DETAILED DESCRIPTION:
The explanation of consciousness poses one of the greatest challenges to science and philosophy in the 21st century. It remains unclear what consciousness is and how it emerges from brain activity. Positron Emission Tomography (PET), Magnetic Resonance Imaging (MRI) and electroencephalography (EEG) studies will be carried out to reveal the neural correlates of consciousness. Consciousness of the subjects will be manipulated with anesthetic agents dexmedetomidine acting through α2-agonism, with propofol and sevoflurane both mainly acting through the enhancement of gamma-aminobutyric acid (GABA) system, and with S-ketamine acting through N-methyl-D-aspartate (NMDA) receptor antagonism. One-hundred-and-sixty (160) healthy male subjects will be recruited to receive EC50 concentration of either dexmedetomidine, propofol, S-ketamine or sevoflurane, or placebo while being imaged for cerebral metabolic rate of glucose (CMRglu). 40 subjects will receive dexmedetomidine, 40 subjects propofol, 20 subjects S-ketamine, 40 subjects sevoflurane and 20 subjects will receive placebo. Also genetic, immunological and metabolomics samples will be taken and analysed to find possible genetic factors explaining the variability in drug response and to find possible immunological and chemical fingerprints of acute drug effect.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age 18-30 years
3. Good general health i.e. American Society of Anesthesiologists (ASA) physical status I
4. Fluent in Finnish language
5. Right handedness
6. Written informed consent
7. Good sleep quality

Exclusion Criteria:

1. Chronic medication
2. History of alcohol and/or drug abuse
3. Strong susceptibility for allergic reactions
4. Serious nausea in connection with previous anesthesia
5. Strong susceptibility for nausea
6. Any use of drugs or alcohol during the 48 hours preceding anesthesia
7. Use of caffeine products 10-12 hours prior the study
8. Smoking
9. Clinically significant previous cardiac arrhythmia / cardiac conduction impairment
10. Clinically significant abnormality in prestudy laboratory tests
11. Positive result in the drug screening test
12. Blood donation within 90 days prior to the study
13. Participation in any medical study with an experimental drug or device during the preceding 60 days
14. The study subject has undergone a prior PET or SPECT study
15. Any contraindication to magnetic resonance imaging (MRI)
16. Hearing impairment
17. Detected unsuitability based on MRI scanning results if available before the PET scanning
18. Sleep disorder or severe sleep problem

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Regional cerebral metabolism of glucose | 40 min
  Comparison of responsive and unresponsive subjects

SECONDARY OUTCOMES:
EEG | 1 hour
  64-channel EEG will be recorded and analyzed using time domain, spectral domain, functional connectivity, directed/effective connectivity and graph theoretical analysis methods.
Immunological effects | 2 hours
  Blood samples will be draw at baseline (without drug), at the end of study drug administration and after PET scanning for the measurement of approximately 50 cytokines, chemokines and growth factors.
Metabolomic effects | 2 hours
  Blood samples will be drawn at baseline (without drug), at the end of drug administration and after PET scanning for the measurement of more than 200 serum measures, including lipoprotein subclass distribution and lipoprotein particle concentration, low molecular weight metabolites, such as amino acids, 3-hydroxybutyrate and creatinine, and detailed molecular information on serum lipids, including free and esterified cholesterol, sphingomyelin and fatty acid saturation.
Gene expression | 2 hours
  Blood samples will be collected at baseline (without drug), at the end of drug administration and after PET scanning for the measurement of RNA expression using whole genome microarray-based, massively parallel sequencing or quantitative reverse-transcription polymerase chain reaction based methods.
Psychological well-being | 2 hours
  Psychological well-being and ill-being will be measured with a battery of scientifically validated scales just before initiating the study session and at the end of the study session.
Dream report | 1 hour
  After terminating PET imaging, a structured interview is immediately conducted to verify a recollection or absence of recollection of subjective experiences during possible loss of responsiveness.

OTHER OUTCOMES:
Drug concentration in plasma or end-tidal | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Harry Scheinin, MD, Principal Investigator — Turku PET Centre, University of Turku, Turku, Finland
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langsjo JW, Alkire MT, Kaskinoro K, Hayama H, Maksimow A, Kaisti KK, Aalto S, Aantaa R, Jaaskelainen SK, Revonsuo A, Scheinin H. Returning from oblivion: imaging the neural core of consciousness. J Neurosci. 2012 Apr 4;32(14):4935-43. doi: 10.1523/JNEUROSCI.4962-11.2012. PMID 22492049
- [Background] Langsjo JW, Revonsuo A, Scheinin H. Harnessing anesthesia and brain imaging for the study of human consciousness. Curr Pharm Des. 2014;20(26):4211-24. PMID 24025060
- [Derived] Nummela A, Laaksonen L, Scheinin A, Kaisti K, Vahlberg T, Neuvonen M, Valli K, Revonsuo A, Perola M, Niemi M, Scheinin H, Laitio T. Circulating oxylipin and bile acid profiles of dexmedetomidine, propofol, sevoflurane, and S-ketamine: a randomised controlled trial using tandem mass spectrometry. BJA Open. 2022 Dec 12;4:100114. doi: 10.1016/j.bjao.2022.100114. eCollection 2022 Dec. PMID 37588789
- [Derived] Nummela AJ, Laaksonen LT, Laitio TT, Kallionpaa RE, Langsjo JW, Scheinin JM, Vahlberg TJ, Koskela HT, Aittomaki V, Valli KJ, Revonsuo A, Niemi M, Perola M, Scheinin H. Effects of dexmedetomidine, propofol, sevoflurane and S-ketamine on the human metabolome: A randomised trial using nuclear magnetic resonance spectroscopy. Eur J Anaesthesiol. 2022 Jun 1;39(6):521-532. doi: 10.1097/EJA.0000000000001591. Epub 2021 Sep 22. PMID 34534172
- [Derived] Laaksonen L, Kallioinen M, Langsjo J, Laitio T, Scheinin A, Scheinin J, Kaisti K, Maksimow A, Kallionpaa RE, Rajala V, Johansson J, Kantonen O, Nyman M, Siren S, Valli K, Revonsuo A, Solin O, Vahlberg T, Alkire M, Scheinin H. Comparative effects of dexmedetomidine, propofol, sevoflurane, and S-ketamine on regional cerebral glucose metabolism in humans: a positron emission tomography study. Br J Anaesth. 2018 Jul;121(1):281-290. doi: 10.1016/j.bja.2018.04.008. Epub 2018 May 8. PMID 29935583